CLINICAL TRIAL: NCT05774678
Title: Trial Of PreoperAtive Radiation (TOPAz): A Randomized Trial Comparing Hypofractionated Versus Conventionally Fractionated Preoperative Radiation Followed by Mastectomy With Immediate Autologous Breast Reconstruction With Integrated Nanomechanical Biomarker Evaluation
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Artidis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-0880; NCI-2023-01985 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2023-02-28; First posted 2023-03-20 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (preoperative radiation hypofractionated) (Experimental): Participants will receive the standard number of radiation treatment doses
  Interventions: Radiation: Group 1 (preoperative radiation hypofractionated); Other: Group 2 (preoperative radiation conventionally fractionated)
- Group 2 (preoperative radiation conventionally fractionated) (Experimental): Participants will receive the standard number of radiation treatment doses
  Interventions: Radiation: Group 1 (preoperative radiation hypofractionated); Other: Group 2 (preoperative radiation conventionally fractionated)

INTERVENTIONS:
Radiation: Group 1 (preoperative radiation hypofractionated) — radiation schedules/regimens before your scheduled breast surgery
Other: Group 2 (preoperative radiation conventionally fractionated) — radiation schedules/regimens before your scheduled breast surgery

SUMMARY:
To compare the outcomes of and responses to 2 different radiation therapy schedules (the standard radiation amount and number of doses versus less radiation and fewer doses) that are being given before having breast cancer surgery (cancer removal and reconstruction).

DETAILED DESCRIPTION:
Primary Objectives:

--To compare BREAST-Q satisfaction with breasts 18 months after reconstructive surgery for patients randomized to HF-PreMRT versus CF-PreMRT. We hypothesize that HF-PreMRT will be superior to CF-PreMRT with regard to this endpoint.

Secondary Objectives:

* To compare oncologic outcomes following HF-PreMRT versus CF-PreMRT, including residual cancer burden, local-regional control, disease-free survival, and overall survival.
* To compare surgical outcomes following HF-PreMRT versus CF-PreMRT, including surgical complications, flap loss, difficulty of reconstructive surgery, number of reoperations, and aesthetic outcomes including photographic assessment of the reconstructed breast.
* To compare radiation outcomes following HF-PreMRT versus CF-PreMRT, including acute and late toxicities and fibrosis.
* To compare health services research outcomes following HF-PreMRT versus CF-PreMRT, including financial toxicity, work productivity and disability, total cost of care, complicationrelated cost of care, and health utility.
* To compare patient-reported quality of life and toxicities following HF-PreMRT versus CFPreMRT.
* To compare patient-reported quality of life and toxicities following HF-PreMRT versus CFPreMRT.
* To evaluate associations between the radiation treatment plan parameters and surgical, radiation, health services, and patient-reported outcomes.
* To evaluate nanomechanical properties of the breast cancer before and after radiation and their association with oncologic outcomes
* To evaluate nanomechanical properties of the breast normal tissue after radiation and their association with surgical and radiation outcomes.
* To evaluate the association of germline polymorphisms, including the pro-fibrotic cytokine transforming growth factor-beta (TGF-β), with circulating serum TGF- levels during and after radiation and toxicities of radiation and reconstruction, particularly fibrotic complications.
* To characterize pre- and post-radiation tumor and nodal tissue by single cell sequencing, whole genome, whole exome, and targeted sequencing, and digital spatial profiling for immune landscape, radiation resistance signatures, microenvironmental and tumor genome profiles and correlate radiation induced changes to tumor and patient characteristics and residual cancer burden.
* To characterize pre- and post-radiation tumor and nodal tissue by single cell sequencing, whole genome, whole exome, and targeted sequencing, and digital spatial profiling for immune landscape, radiation resistance signatures, microenvironmental and tumor genome profiles and correlate radiation induced changes to tumor and patient characteristics and residual cancer burden.
* To characterize irradiated normal breast and nodal tissues for genomic, proteomic, and metabolomic profiles and correlate these to tumor and patient characteristics, tumor burden, and toxicity
* To characterize irradiated normal breast and nodal tissues for genomic, proteomic, and metabolomic profiles and correlate these to tumor and patient characteristics, tumor burden, and toxicity.
* To compare surgical, radiation, and health services outcomes for patients treated with PreMRT on this trial to a matched cohort of patients treated with standard post-mastectomy radiation with breast reconstruction on the SAPHIRE protocol (2016-0142).
* To compare translational data for patients treated with PreMRT on this trial to a matched cohort of patients treated with standard post-mastectomy radiation with breast reconstruction on the SAPHIRE protocol (2016-0142).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Histologic diagnosis of invasive breast cancer (cytologic or histologic confirmation of nodal metastasis is sufficient to establish this eligibility criteria).
* Clinical and/or pathologic stage T3-T4c OR N1-N3; for the IBC pilot cohort only, the stage requirement is T4d, any N, M1
* Mastectomy is the planned oncologic surgery but has not yet been performed at the time of protocol enrollment
* Autologous (i.e. tissue-based) reconstruction is planned with either a free or rotational flap.
* For patients with HER2 positive, non-IBC breast cancer treated with neoadjuvant chemotherapy, one of the following criteria must be met:

  1. Residual invasive disease should be documented in either the breast or a regional nodal metastasis after neoadjuvant chemotherapy. This specific eligibility criteria can be satisfied by the post-chemotherapy standard of care breast biopsy. For this matter, the patient may be enrolled on the trial prior to biopsy. If the biopsy does not show residual invasive disease, then the patient will not proceed with protocol-directed therapy and will be removed and replaced from the study.
  2. Medical oncologist has documented a discussion in the chart about potential risks of proceeding with PreMRT with regard to impact on adjuvant systemic therapy decisions and the patient has opted to proceed with trial enrollment
* For T4d pilot cohort patients, post-chemotherapy, pre-radiation ultrasound must demonstrate at least partial response in the breast and regional lymph nodes and no suspicious infraclavicular, internal mammary, and supraclavicular lymph nodes.
* Ability to provide written informed consent in accordance with institutional policies.

Exclusion Criteria:

* Patients undergoing treatment for recurrent breast cancer in the index breast or lymph nodes.
* History of therapeutic irradiation to the breast, lower neck, mediastinum or other area(s) that will overlap with the affected breast.
* Presence of active scleroderma
* Patients who are pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2023-04-05 (Actual); Primary Completion 2026-11-01 (Estimated); Study Completion 2028-11-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version (v) 5.0 | through study completion; an average of 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D. Smith, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Schaverien MV, Singh P, Kuerer HM, Akay CL, Chavez-MacGregor M, Chu CK, Clemens MW, Qiao W, Smith BD, Hoffman KE. Comparison of Outcomes of Microsurgical Breast Reconstruction after Premastectomy and Postmastectomy Radiation Therapy. J Am Coll Surg. 2025 Oct 1;241(4):535-549. doi: 10.1097/XCS.0000000000001444. Epub 2025 Sep 16. PMID 40366003
- [Derived] Schaverien MV, Singh P, Smith BD, Qiao W, Akay CL, Bloom ES, Chavez-MacGregor M, Chu CK, Clemens MW, Colen JS, Ehlers RA, Hwang RF, Joyner MM, Largo RD, Mericli AF, Mitchell MP, Shuck JW, Tamirisa N, Tripathy D, Villa MT, Woodward WA, Zacharia R, Kuerer HM, Hoffman KE. Premastectomy Radiotherapy and Immediate Breast Reconstruction: A Randomized Clinical Trial. JAMA Netw Open. 2024 Apr 1;7(4):e245217. doi: 10.1001/jamanetworkopen.2024.5217. PMID 38578640
- See also: M D Anderson Cancer Center — http://www.mdanderson.org